CLINICAL TRIAL: NCT01539928
Title: Dual PET/CT Imaging in Lung Cancer (Danish Title: En og Tre Timers FDG-PET/CT Ved Lungecancer)
Brief Title: Dual PET/CT Imaging in Lung Cancer
Acronym: DILUCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mie Holm Vilstrup, Principal investigator, MD, Odense University Hospital
Other Study IDs: NMA 61 DILUCE
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: Dual time PET/CT; glucose-6-phosphatase
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh frozen sample of primary lung cancer tumor
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lung cancer or high suspicion of lung cancer: After initial work-up (chest x-ray, CT of thorax and upper abdomen, spirometry) found to have surgically resectable lung cancer
  Interventions: Other: Dual FDG-PET/CT

INTERVENTIONS:
Other: Dual FDG-PET/CT — Conventional FDG-PET/CT preformed after 1 hour and additional PET/CT 3 hours after injection

SUMMARY:
The purpose of this study is to compare conventional PET/CT scan performed 1 hour after injection of the radioactive tracer FDG (PET/CT[1]) with PET/CT performed after 3 hours (PET/CT[3]) in a group of patients with biopsy verified lung cancer or high suspicion of lung cancer after initial work-up (chest x-ray and CT of thorax/upper abdomen), who are potentially operable.

DETAILED DESCRIPTION:
The investigators also want to:

* To find the sensitivity, specificity and accuracy in PET/CT 1h and 3 h in the staging of lung cancer (N-/M-stage). Our gold standard is pathology, when not possible - follow-up (se Gold Standard 6.1.1)
* To compare SUVmax with the expression of GLUT1 and G-6-Pase in tumors
* To compare the expression of GLUT1 with the activity of G6Pase
* To compare SUVmax, RI, tumor/liver ratio, GLUT1 and G-6-Pase with the occurrence of relapse within a year after curative surgery

ELIGIBILITY:
Inclusion Criteria:

* Cytologic/histologic-verified lung cancer or high suspicion of lung cancer after initial work up
* Candidate to curative intended surgery after initial work up (usually chest x-ray, CT of chest/upper abdomen and if needed spirometry).

Exclusion Criteria:

* Former lung cancer
* Contraindications for PET/CT: Pregnancy, recent chemoradiotherapy
* Diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pt. referred to The Department of Pulmonary Medicine, Odense University Hospital or The Department of Medicine, Hospital of Southern Denmark, Sønderborg with suspicion of lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity and accuracy | After staging or 1 year of follow up
  To find the sensitivity, specificity and accuracy in PET/CT 1h and 3 h in the staging of lung cancer (N-/M-stage). Our gold standard is pathology, when not possible - follow-up

SECONDARY OUTCOMES:
Occurence of relapse | 1 year follow up after surgery
  • To compare SUVmax, RI, tumor/liver ratio, GLUT1 and G-6-Pase with the occurrence of relapse within a year after curative surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mie H Vilstrup, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Pulmonary Medicine, Odense C, Fünen, Denmark